CLINICAL TRIAL: NCT00796068
Title: Transplantation of Umbilical Cord Blood in Patients With Hematological Malignancies Using a Treosulfan Based Preparative Regimen
Brief Title: Treosulfan, Fludarabine Phosphate, and Total-Body Irradiation in Treating Patients With Hematological Cancer Who Are Undergoing Umbilical Cord Blood Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Principal Investigator, Filippo Milano, Associate Professor, Fred Hutchinson Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2275.00; NCI-2010-00299 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2275; 2275.00 (Other: Fred Hutch/University of Washington Cancer Consortium); RG2808000 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Results first posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-01

CONDITIONS: Acute Biphenotypic Leukemia; Acute Lymphoblastic Leukemia in Remission; Acute Myeloid Leukemia in Remission; Blasts Under 5 Percent of Bone Marrow Nucleated Cells; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Chronic Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Myelodysplastic Syndrome (MDS)
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase; Myelodysplastic Syndromes | interventions — Cyclosporine; Cyclosporins; fludarabine phosphate; Mycophenolic Acid; Whole-Body Irradiation; treosulfan; Cord Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (low risk for graft failure) (Experimental): Patients receive a conditioning regimen comprising fludarabine phosphate IV over 1 hour QD on days -6 to -2 and treosulfan IV over 120 minutes on days - 6 to -4. Patients undergo TBI on day -1. Patients then undergo donor UCBT on day 0.
  Patients receive GVHD prophylaxis comprising cyclosporine IV over 1 hour or PO 2-3 times daily on days -3 to 100, followed by a taper in the absence of GVHD. Patients also receive mycophenolate mofetil IV 3 times daily on days 0 to 40, followed by a taper in the absence of GVHD.
  Interventions: Drug: Cyclosporine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Radiation: Total-Body Irradiation; Drug: Treosulfan; Procedure: Umbilical Cord Blood Transplantation
- Arm II (high risk for graft failure) (Experimental): Patients receive a conditioning regimen, TBI, donor UCBT, GVHD prophylaxis, and mycophenolate mofetil as in Arm I.
  Interventions: Drug: Cyclosporine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Radiation: Total-Body Irradiation; Drug: Treosulfan; Procedure: Umbilical Cord Blood Transplantation

INTERVENTIONS:
Drug: Cyclosporine — Given IV or PO
  Other Names: 27-400; Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Gengraf; Neoral; OL 27-400; Sandimmun; Sandimmune; SangCya
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mycophenolate Mofetil — Given IV
  Other Names: Cellcept; MMF
Radiation: Total-Body Irradiation — TBI administered day -1: 200 cGy (or escalated to 300 cGy, 400 cGy, or 450 cGy per protocol statistical section)
  Other Names: Total Body Irradiation; Whole-Body Irradiation
Drug: Treosulfan — Given IV
  Other Names: 1,2,3, 4-Butanetetrol, 1,4-dimethanesulfonate, [R-(R*,S*)]-; Dihydroxybusulfan; Ovastat; Treosulphan; Tresulfon
Procedure: Umbilical Cord Blood Transplantation — Undergo single or double unit UCBT
  Other Names: Cord Blood Transplantation; UCB transplantation

SUMMARY:
This phase II trial studies how well giving treosulfan together with fludarabine phosphate and total-body irradiation (TBI) works in treating patients with hematological cancer who are undergoing umbilical cord blood transplant (UCBT). Giving chemotherapy, such as treosulfan and fludarabine phosphate, and TBI before a donor UCBT helps stop the growth of cancer cells and helps stop the patient's immune system from rejecting the donor's stem cells. When the stem cells from a related or unrelated donor, that do not exactly match the patient's blood, are infused into the patient, they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine (CsA) and mycophenolate mofetil (MMF) after the transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Graft failure/rejection and secondary graft failure.

II. Day -200 non-relapse mortality.

SECONDARY OBJECTIVES:

I. Platelet engraftment by six months.

II. Grade II-IV and III-IV acute graft-versus-host disease (GVHD) at day 100 and one year.

III. Chronic GVHD.

IV. Clinically significant infections.

V. Overall survival.

VI. Relapse or disease progression.

VII. Immune reconstitution (Fred Hutchinson Cancer Research Center [FHCRC] only).

VIII. Emergence of a dominant unit (FHCRC only).

OUTLINE: Patients are assigned to 1 of 2 arms.

ARM I (low risk for graft failure): Patients receive a conditioning regimen comprising fludarabine phosphate intravenously (IV) over 1 hour once daily (QD) on days -6 to -2 and treosulfan IV over 120 minutes on days - 6 to -4. Patients undergo TBI on day -1. Patients then undergo donor UCBT on day 0. Patients receive GVHD prophylaxis comprising cyclosporine IV over 1 hour or orally (PO) 2-3 times daily on days -3 to 100, followed by a taper in the absence of GVHD. Patients also receive mycophenolate mofetil IV 3 times daily on days 0 to 40, followed by a taper in the absence of GVHD.

ARM II (high risk for graft failure): Patients receive a conditioning regimen, TBI, donor UCBT, GVHD prophylaxis, and mycophenolate mofetil as in Arm I.

After completion of the study treatment, patients are followed up at 6 months and 1 and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Acute myeloid leukemia/acute lymphoblastic leukemia, including biphenotypic acute leukemia or mixed-lineage leukemia: Must have < 5% morphologic marrow blasts in an evaluable marrow sample (> 25% of normal cellularity for age collected less than one month prior to start of conditioning; patients in which adequate marrow/biopsy specimens cannot be obtained to determine remission status by morphologic assessment, but have fulfilled criteria of remission by flow cytometry, recovery of peripheral blood counts with no circulating blasts, and/or normal cytogenetics (if applicable) may still be eligible; reasonable attempts must be made to obtain an adequate specimen for morphologic assessment, including possible repeat procedures; these patients must be discussed with the principal investigator prior to enrollment; patients persistently aplastic for greater than one month since completing last chemotherapy are also eligible with principal investigator (PI) approval
* Myelodysplastic syndrome (MDS): Any 2001 World Health Organization (WHO) classification subtype; refractory anemia with excess blasts (RAEB)-2 patients may proceed directly to transplant, but may also be considered for induction chemotherapy before transplant; patients with >= 20% morphologic marrow blasts require induction therapy to reduce morphologic marrow blasts below 5% before transplant
* Chronic myelogenous leukemia: All types, except refractory blast crisis; chronic phase patients must have failed or been intolerant to Gleevec or other tyrosine kinase inhibitors
* Patients =< 50 must have performance status score: Karnofsky (for adults) >= 70 or Eastern Cooperative Oncology Group (ECOG) 0-1; Lansky (for children) score >= 50
* Patients > 50 must have Karnofsky performance score >= 70 or ECOG 0-1 and comorbidity index < 5
* Adequate cardiac function defined as absence of decompensated congestive heart failure or uncontrolled arrhythmia AND left ventricular ejection fraction >= 35% OR fractional shortening > 22%
* Adequate pulmonary function defined as absence of oxygen (O2) requirements and one of the following:

  * Diffusion lung capacity for carbon monoxide (DLCO) corrected >= 70% mm Hg
  * DLCO corrected between 60% - 69% mm Hg and partial pressure of oxygen (pO2) >= 70 mm Hg
  * DLCO corrected between 50% - 59% mm Hg and pO2 >= 80 mm Hg
  * Pediatric patients unable to perform pulmonary function tests must have O2 saturation > 92% on room air; may not be on supplemental oxygen
* Adequate hepatic function; patients with clinical or laboratory evidence of liver disease will be evaluated for the cause of liver disease, its clinical severity in terms of liver function, histology, and the degree of portal hypertension; patients with fulminant liver failure, cirrhosis with evidence of portal hypertension or bridging fibrosis, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, or correctable hepatic synthetic dysfunction evidenced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3 mg/dL, and symptomatic biliary disease will be excluded
* Adequate renal function defined as creatinine =< 2.0 mg/dl (adults) or estimated creatinine clearance > 40 ml/min (pediatrics); all adults with a creatinine > 1.2 or a history of renal dysfunction must have estimated creatinine clearance > 40 ml/min
* If recent mold infection, e.g., Aspergillus, must be cleared by infectious disease to proceed
* Prior hematopoietic cell transplant: must be >= 3 months after previous transplant
* DONOR: Human leukocyte antigen (HLA) matching:

  * Minimum requirement: The cord blood (CB) graft(s) must be matched at a minimum at 4/6 HLA-A, B, DRB1 loci with the recipient; therefore 0-2 mismatches at the A or B or DRB1 loci based on intermediate resolution A, B antigen and DRB1 allele typing for determination of HLA-match is allowed
  * HLA-matching determined by high resolution typing is allowed per institutional guidelines as long as the minimum criteria (above) are met
* DONOR: Selection of two CB units is mandatory when a single cord blood unit does not meet the following criteria in the table below

  * Match grade

    * 6/6

      * Single unit allowed for total nucleated cell (TNC) dose >= 2.5 x 10^7/kg
    * 5/6, 4/6

      * Single unit allowed for TNC dose >= 4.0 (+/- 0.5) x 10^7/kg
  * If two CB units are used, the total cell dose of the combined units must be at least 3.0 x 10^7 TNC per kilogram recipient weight based on pre-cryopreservation numbers, with each CB unit containing a MINIMUM of 1.5 x 10^7 TNC/kg
* DONOR: The minimum recommended CD34/kg cell dose should be 2 x 10^5 CD34/kg, total dose from a single or combined double
* DONOR: The unmanipulated CB unit(s) will be Food and Drug Administration (FDA) licensed or will be obtained under a separate investigational new drug (IND), such as the National Marrow Donor Program (NMDP) Protocol 10-CBA conducted under BB IND-7555 or another IND sponsored by (1) a participating institution or (2) an investigator at FHCRC or one of the participating institutions
* DONOR (FHCRC only): Up to 5% of the unmanipulated cord blood product (s), when ready for infusion, may be withheld for research purposes as long as thresholds for infused TNC dose are met; these products will be used to conduct studies involving the kinetics of engraftment and immunobiology of double cord transplantation

Exclusion Criteria:

* Pregnancy or breastfeeding
* Evidence of human immunodeficiency virus (HIV) infection or known HIV positive serology
* Uncontrolled viral or bacterial infection at the time of study enrollment
* Active or recent (prior 6 month) invasive fungal infection without infectious diseases (ID) consult and approval
* Central nervous system (CNS) leukemic involvement not clearing with intrathecal chemotherapy and/or cranial radiation prior to initiation of conditioning (day -6)
* DONOR: Any cord blood units with < 1.5 x 10^7 total nucleated cells per kilogram recipient weight
* DONOR: Any cord blood units that have not passed donor screening for infectious disease markers as recommended by NMDP will not be used unless a waiver is signed by the clinical attending allowing use of CB unit. Cord blood units are presumed to be cytomegalovirus (CMV) negative regardless of serologic testing due to passive transmission of maternal CMV antibodies

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2009-02-24 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Milano, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (3):
- United States (3):
  - University of Colorado Hospital, Aurora, Colorado
  - Oregon Health and Science University, Portland, Oregon
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

REFERENCES:
- [Derived] Milano F, Gutman JA, Deeg HJ, Nemecek ER, Baumgart J, Thur L, Dahlberg A, Salit RB, Summers C, Appelbaum FR, Delaney C. Treosulfan-based conditioning is feasible and effective for cord blood recipients: a phase 2 multicenter study. Blood Adv. 2020 Jul 28;4(14):3302-3310. doi: 10.1182/bloodadvances.2020002222. PMID 32706891

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between February 2009 and October 2019, 130 cord blood transplant (CBT) recipients were enrolled in this prospective multi-center phase II study.
Pre-assignment Details: All participants who signed consent were assigned to one of two arms and all completed enrollment.
Groups:
- Arm I (Low Risk for Graft Failure): Patients receive a conditioning regimen comprising fludarabine phosphate intravenously (IV) over 1 hour every day (QD) on days -6 to -2 and treosulfan IV over 120 minutes on days - 6 to -4. Patients undergo total body irradiation (TBI) on day -1. Patients then undergo donor cord blood transplant (CBT) on day 0.
  Patients receive graft versus host disease (GVHD) prophylaxis comprising cyclosporine IV over 1 hour or by mouth (PO) 2-3 times daily on days -3 to 100, followed by a taper in the absence of GVHD. Patients also receive mycophenolate mofetil IV 3 times daily on days 0 to 40, followed by a taper in the absence of GVHD.
  Cyclosporine: Given IV or PO
  Fludarabine Phosphate: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Mycophenolate Mofetil: Given IV
  Total-Body Irradiation: TBI administered day -1: 200 centigray (cGy) (or escalated to 300 cGy, 400 cGy, or 450 cGy per protocol statistical section)
  Treosulfan: Given IV
  Umbilical Cord Blood Transplantation (UCBT): Undergo single or double unit UCBT
- Arm II (High Risk for Graft Failure): Patients receive a conditioning regimen, total body irradiation (TBI), donor cord blood transplant (CBT), graft versus host disease (GVHD) prophylaxis, and mycophenolate mofetil as in Arm I.
  Cyclosporine: Given intravenously (IV) or by mouth (PO)
  Fludarabine Phosphate: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Mycophenolate Mofetil: Given IV
  Total-Body Irradiation: TBI administered day -1: 200 centigray (cGy) (or escalated to 300 cGy, 400 cGy, or 450 cGy per protocol statistical section)
  Treosulfan: Given IV
  Umbilical Cord Blood Transplantation (UCBT): Undergo single or double unit UCBT
Period: Overall Study
Arm/Group | Arm I (Low Risk for Graft Failure) | Arm II (High Risk for Graft Failure)
Started | 66 | 64
Completed | 66 | 64
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm I (Low Risk for Graft Failure): Patients receive a conditioning regimen comprising fludarabine phosphate IV over 1 hour every day (QD) on days -6 to -2 and treosulfan IV over 120 minutes on days - 6 to -4. Patients undergo total body irradiation (TBI) on day -1. Patients then undergo donor umbilical cord blood transplantation (UCBT) on day 0.
  Patients receive graft-versus-host disease (GVHD) prophylaxis comprising cyclosporine IV over 1 hour or by mouth (PO) 2-3 times daily on days -3 to 100, followed by a taper in the absence of GVHD. Patients also receive mycophenolate mofetil IV 3 times daily on days 0 to 40, followed by a taper in the absence of GVHD.
  Cyclosporine: Given IV or PO
  Fludarabine Phosphate: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Mycophenolate Mofetil (MMF): Given IV
  Total-Body Irradiation: TBI administered day -1: 200 cGy (or escalated to 300 cGy, 400 cGy, or 450 cGy per protocol statistical section)
  Treosulfan: Given IV
  Umbilical Cord Blood Transplantation: Undergo single or double unit UCBT
- Total: Total of all reporting groups
Arm/Group | Arm I (Low Risk for Graft Failure) | Arm II (High Risk for Graft Failure) | Total
Number analyzed (Participants) | 66 | 64 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18 | 13 | 31
  Between 18 and 65 years | 46 | 51 | 97
  >=65 years | 2 | 0 | 2
Age, Continuous [Median (Full Range); unit: years] | 47 [0.6 to 65] | 43 [2 to 64] | 45 [0.6 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 33 | 69
  Male | 30 | 31 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants] — Racial and ethnicity categories based on the Office of Management and Budget (OMB) and the National Institutes of Health (NIH) minimum categories for race and ethnicity.
  Participants
    American Indian or Alaska Native | 1 | 2 | 3
    Asian | 7 | 12 | 19
    Native Hawaiian or Other Pacific Islander | 4 | 4 | 8
    Black or African American | 1 | 4 | 5
    White | 38 | 36 | 74
    More than one race | 2 | 1 | 3
    Unknown or Not Reported | 13 | 5 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 66 | 64 | 130
Hematopoietic Cell Transplantation-Comorbidity Index (HCT-CI) [Median (Full Range); unit: units on a scale] — Hematopoietic Cell Transplantation-Comorbidity Index (HCT-CI). The HCT-CI is a comorbidity index that comprises 17 different categories of organ dysfunction. Positive findings are summated into a total score. The HCT-CI provides information with regard to the overall as well as non-relapse mortality risk a patient is likely to experience after hematopoietic cell transplantation. The HCT-CI scores were further collapsed into 3 risk groups: . A score of 0 indicates low risk, a score of 1-2 indicates intermediate risk and any score ≥3 indicates a high risk of non-relapse mortality.
  units on a scale | 2 [0 to 5] | 2 [0 to 6] | 2 [0 to 6]
Diagnosis [Count of Participants; unit: Participants]
  Acute myeloid leukemia (AML) | 38 | 25 | 63
  Acute lymphoblastic leukemia (ALL) | 24 | 13 | 37
  Biphenotypic | 1 | 1 | 2
  Myelodysplastic Syndrome (MDS) | 3 | 22 | 25
  Myeloproliferative | 0 | 3 | 3
Human leukocyte antigens (HLA) matching to recipients [Count of Participants; unit: Participants] — A close match between a donor's and a patient's HLA markers is essential for a successful transplant outcome. HLA matching promotes the growth and development of new healthy blood cells (called engraftment) and reduces the risk of a post-transplant complication called graft-versus-host (GVHD) disease.
  Participants
    6/6 | 3 | 2 | 5
    5/6 | 25 | 17 | 42
    4/6 | 38 | 45 | 83

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Graft Failure/Rejection
Description: Patients will be considered primary graft failure provided they meet any criteria listed below, in the absence of documented disease persistence/recurrence or active bone marrow infection (ex. Cytomegalovirus (CMV)):
  i. Absence of 3 consecutive days with neutrophils >500/u1 combined with host CD3+ peripheral blood chimerism ≥50% at day 42 ii. Absence of 3 consecutive days with neutrophils >500/u1 under any circumstances at day 55 iii. Death after day 28 with neutrophil count <100/u1 without any evidence of engraftment (< 5% donor CD3+) iv. Primary autologous count recovery with < 5% donor CD3+ peripheral blood chimerism at count recovery and without relapse
Time Frame: Up to 100 days
Measure: Count of Participants; unit: Participants
Groups:
- Arm I (Low Risk for Graft Failure): Patients receive a conditioning regimen comprising fludarabine phosphate IV over 1 hour QD on days -6 to -2 and treosulfan IV over 120 minutes on days - 6 to -4. Patients undergo TBI on day -1. Patients then undergo donor UCBT on day 0.
  Patients receive GVHD prophylaxis comprising cyclosporine IV over 1 hour or PO 2-3 times daily on days -3 to 100, followed by a taper in the absence of GVHD. Patients also receive mycophenolate mofetil IV 3 times daily on days 0 to 40, followed by a taper in the absence of GVHD.
  Cyclosporine: Given IV or PO
  Fludarabine Phosphate: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Mycophenolate Mofetil: Given IV
  Total-Body Irradiation: TBI administered day -1: 200 cGy (or escalated to 300 cGy, 400 cGy, or 450 cGy per protocol statistical section)
  Treosulfan: Given IV
  Umbilical Cord Blood Transplantation: Undergo single or double unit UCBT
Arm/Group | Arm I (Low Risk for Graft Failure) | Arm II (High Risk for Graft Failure)
Number analyzed (Participants) | 66 | 64
Participants | 2 | 5

2. Primary Outcome: Number of Participants With Secondary Graft Failure
Description: Secondary graft failure is defined as decline of neutrophil count to <500/ul with loss of donor chimerism after day 55
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Low Risk for Graft Failure) | Arm II (High Risk for Graft Failure)
Number analyzed (Participants) | 66 | 64
Participants | 0 | 0

3. Primary Outcome: Number of Patients With Non-relapse Mortality (NRM)
Description: Defined as death from any cause without sign of disease progression or relapse. Loss to follow up are censored, whereas disease relapse or progression are considered competing risks.
Time Frame: At day -200
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Low Risk for Graft Failure) | Arm II (High Risk for Graft Failure)
Number analyzed (Participants) | 66 | 64
Participants | 7 | 6

4. Secondary Outcome: Number of Participants Surviving by 1 Year
Description: Overall survival was measured from the first day of CBT infusion until death from any cause.
Time Frame: At 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Low Risk for Graft Failure) | Arm II (High Risk for Graft Failure)
Number analyzed (Participants) | 66 | 64
Participants | 51 | 47

5. Secondary Outcome: The Number of Participants Alive at Two-years Follow up.
Description: Overall survival of participants after two-years of follow up.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Low Risk for Graft Failure) | Arm II (High Risk for Graft Failure)
Number analyzed (Participants) | 66 | 64
Participants | 50 | 44

6. Secondary Outcome: Non-relapse Mortality
Description: Death of any cause other than relapse or disease progression was considered.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Low Risk for Graft Failure) | Arm II (High Risk for Graft Failure)
Number analyzed (Participants) | 66 | 64
Participants | 8 | 10

7. Secondary Outcome: Duration (Days) Until Participants Obtained Platelet Engraftment
Description: Summarized using a range and median of measure in days until participants reached platelet engraftment. Platelet engraftment was defined as the first of 7 consecutive days when the platelet count exceeded 20 x 109/L (untransfused).
Time Frame: At 6 months
Measure: Median (Full Range); unit: days
Arm/Group | Arm I (Low Risk for Graft Failure) | Arm II (High Risk for Graft Failure)
Number analyzed (Participants) | 66 | 64
days | 31 [16 to 83] | 31 [12 to 87]

8. Secondary Outcome: Number of Participants With Acute Graft-versus-host Disease (GVHD) Grade II-IV by Day 100
Description: Grade I GVHD is characterized as mild disease, grade II GVHD as moderate, grade III as severe, and grade IV life-threatening. Diagnosing and grading acute GVHD is based on clinical findings (the organ stage, response to treatment and whether GVHD was a major cause of death) and frequently varies between transplant centers and independent reviewers.
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Low Risk for Graft Failure) | Arm II (High Risk for Graft Failure)
Number analyzed (Participants) | 66 | 64
Participants | 36 | 37

9. Secondary Outcome: Incidence of Acute or Chronic Graft-versus-host Disease (GVHD)
Description: Overall GVHD is determined based on the organ stage, response to treatment and whether GVHD was a major cause of death. Chronic GVHD will be defined according to the National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease. Described as mild, moderate, or severe as graded according to the attached Organ Scoring Sheet. Symptoms consistent with both chronic and acute GVHD occurring after day 100 will be considered overlap chronic GVHD syndrome.
Time Frame: At 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Low Risk for Graft Failure) | Arm II (High Risk for Graft Failure)
Number analyzed (Participants) | 66 | 64
Participants | 7 | 6

10. Secondary Outcome: Incidence of Relapse or Disease Progression
Description: Cumulative incidence estimates using non-relapse mortality as competitive event.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Low Risk for Graft Failure) | Arm II (High Risk for Graft Failure)
Number analyzed (Participants) | 66 | 64
Participants | 17 | 11

11. Secondary Outcome: Number of Participants Surviving up to 2 Years Without Disease Progression
Description: Progression-free survival is the time interval from start of treatment to documented evidence of disease progression. Disease progression was defined by European LeukemiaNet 2017 criteria and International Working Group (IWG) within 3 years of transplant.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Low Risk for Graft Failure) | Arm II (High Risk for Graft Failure)
Number analyzed (Participants) | 66 | 64
Participants | 37 | 41

12. Secondary Outcome: Incidence of Clinically Significant Infections
Description: Collected and graded according to the modified National Cancer Institute Common Toxicity Criteria.
Time Frame: At 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Low Risk for Graft Failure) | Arm II (High Risk for Graft Failure)
Number analyzed (Participants) | 66 | 64
Participants | 53 | 61

ADVERSE EVENTS:
Time Frame: Adverse events (AE) will be monitored and recorded in study-specific case report forms (CRFs) from the time of first exposure to an investigational product in this study through day +100 post-transplant. The start of the adverse event reporting for a study subject will coincide with signing of the informed consent. All-cause mortality data was censored at two-year follow-up.
Groups:
- Arm I (Low Risk for Graft Failure): Patients receive a conditioning regimen comprising fludarabine phosphate IV over 1 hour every day (QD) on days -6 to -2 and treosulfan IV over 120 minutes on days - 6 to -4. Patients undergo (total body irradiation (TBI) on day -1. Patients then undergo donor cord blood transplantation (CBT) on day 0.
  Patients receive graft-versus-host disease (GVHD) prophylaxis comprising cyclosporine IV over 1 hour or by mouth (PO) 2-3 times daily on days -3 to 100, followed by a taper in the absence of GVHD. Patients also receive mycophenolate mofetil IV 3 times daily on days 0 to 40, followed by a taper in the absence of GVHD.
  Cyclosporine: Given IV or PO
  Fludarabine Phosphate: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Mycophenolate Mofetil: Given IV
  Total-Body Irradiation: TBI administered day -1: 200 centigray (cGy) (or escalated to 300 cGy, 400 cGy, or 450 cGy per protocol statistical section)
  Treosulfan: Given IV
  Umbilical Cord Blood Transplantation (UCBT): Undergo single or double unit UCBT
Arm/Group | Arm I (Low Risk for Graft Failure) | Arm II (High Risk for Graft Failure)
All-Cause Mortality (participants affected / at risk) | 16/66 | 20/64
Serious Adverse Events (participants affected / at risk) | 27/66 | 23/64
Other Adverse Events (participants affected / at risk) | 63/66 | 59/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Low Risk for Graft Failure) (N=66) | Arm II (High Risk for Graft Failure) (N=64)
Allergic Reaction (Immune system disorders) | 0 (0) | 1 (1)
Acute cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Left Ventricular Systolic dysfunction (Cardiac disorders) | 3 (3) | 1 (1)
Cardiac troponin I increased (Investigations) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 2 (2) | 0 (0)
Infusional Toxicity/Stunned Heart (Cardiac disorders) | 0 (0) | 1 (1)
Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Sinusoidal obstruction syndrome (Hepatobiliary disorders) | 0 (0) | 2 (2)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 2 (2)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Myelitis (Infections and infestations) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 2 (3) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Other - autonomic dysreflexia exacerbation (Nervous system disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 3 (3)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Anorectal infection (Infections and infestations) | 1 (1) | 0 (0)
Encephalitis infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Low Risk for Graft Failure) (N=66) | Arm II (High Risk for Graft Failure) (N=64)
Allergic Reaction (Immune system disorders) | 2 (2) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Flutter (Cardiac disorders) | 2 (2) | 0
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 11 (11) | 10 (10)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Disemminated vascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Sinusoidal obstruction syndrome (Hepatobiliary disorders) | 1 (1) | 0 (0)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 13 (13) | 6 (6)
Colitis (Gastrointestinal disorders) | 3 (3) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 0 (0)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis (Gastrointestinal disorders) | 10 (10) | 11 (11)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 11 (11) | 12 (12)
Febrile Neutropenia (Blood and lymphatic system disorders) | 27 (27) | 28 (28)
Sepsis (Infections and infestations) | 25 (33) | 31 (45)
Lung infection (Infections and infestations) | 4 (4) | 4 (6)
Urinary tract infection (Infections and infestations) | 5 (6) | 7 (7)
Skin infection (Infections and infestations) | 2 (2) | 5 (6)
Encephalitis infection (Infections and infestations) | 2 (2) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 4 (4) | 3 (3)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 3 (3) | 5 (5)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 18 (19)
Creatinine increased (Investigations) | 2 (2) | 5 (5)
Renal failure (Renal and urinary disorders) | 1 (1) | 4 (4)
Left Ventricular Systolic dysfunction (Cardiac disorders) | 0 (0) | 9 (9)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 0 (0) | 2 (2)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Gatritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Otitis Externa (Infections and infestations) | 0 (0) | 1 (1)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Duodenal infection (Infections and infestations) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Oral cavity (Infections and infestations) | 2 (2) | 0 (0)
Other: genitourinary (Infections and infestations) | 4 (5) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Anorectal infection (Infections and infestations) | 1 (1) | 0 (0)
Other: pulmonary insufficiency (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Other: Thrombosis (Vascular disorders) | 3 (3) | 2 (2)
Other: Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Other: Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Other: Genitalia infection (Infections and infestations) | 1 (1) | 0 (0)
Other: Melena (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/68/NCT00796068/Prot_SAP_000.pdf